CLINICAL TRIAL: NCT00907881
Title: Prospective Observational Study to Assess Correlation Between Glycemic Control and Hypoglycemia in Patients With Type 2 Diabetes Treated With Sulfonylurea
Brief Title: The OBSTACLE Hypoglycemia Study (MK-0000-158)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0000-158; 2009_001
Record Dates: First submitted 2009-05-21; First posted 2009-05-25 (Estimated); Results first posted 2011-11-24 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sulfonylurea Compounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- All participants: Participants with type 2 diabetes mellitus (T2DM) who had sulfonylurea treatment added to an on-going regime of oral hypoglycemic agent(s).
  Interventions: Drug: Sulfonylurea

INTERVENTIONS:
Drug: Sulfonylurea — The dose and frequency of administration of study drug (sulfonylurea) was decided by the investigator according to the individual need of each participant.

SUMMARY:
This study will assess the correlation between glycemic control and the hypoglycemia symptom score in patients with Type 2 diabetes, 12 weeks after addition of a sulfonylurea to an ongoing regime of oral hypoglycemic agents.

DETAILED DESCRIPTION:
Patients will be evaluated for participation in the study during their usual visit to participating diabetes care clinics. Addition of sulfonylurea will be an unbiased decision of the participating physicians based on the clinical needs of the participating patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 Diabetes, of either gender and aged between 18-75 years
* Patients being considered for addition of Sulfonylurea on background of at least one other oral hypoglycemic agent, on a usual visit (screening cum enrolment visit), as per the clinical situation judged by participating physician
* Willing to comply with study requirements

Exclusion Criteria:

* Patients with type 1 Diabetes or gestational Diabetes
* Patients currently on insulin therapy or have received Insulin in last 6 months
* Patients currently on Sulfonylurea therapy or have received Sulfonylureas in last 6 months
* Patients currently on Meglitinides therapy or have received Meglitinides in last 6 months
* Patients initiated on Sulfonylurea monotherapy
* Patient on DPP-4 inhibitors, either as monotherapy or as combination therapy
* Patient is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Patients for whom it would be impossible to complete the questionnaire for whatever reason, in any feasible form
* Patients who are already participating in a clinical trial or other clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 1069 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Kalra S, Deepak MC, Narang P, Singh V, Uvaraj MG, Agrawal N. Usage pattern, glycemic improvement, hypoglycemia, and body mass index changes with sulfonylureas in real-life clinical practice: results from OBSTACLE Hypoglycemia Study. Diabetes Technol Ther. 2013 Feb;15(2):129-35. doi: 10.1089/dia.2012.0237. Epub 2013 Jan 5. PMID 23289432
- [Derived] Kalra S, Deepak MC, Narang P, Singh V, Maheshwari A. Correlation between measures of hypoglycemia and glycemic improvement in sulfonylurea treated patients with type 2 diabetes in India: results from the OBSTACLE hypoglycemia study. J Postgrad Med. 2014 Apr-Jun;60(2):151-5. doi: 10.4103/0022-3859.132322. PMID 24823514

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 1069
Completed | 984
Not Completed | 85
Not completed — Lost to Follow-up | 59
Not completed — Noncompliance | 5
Not completed — Withdrawal by Subject | 5
Not completed — Protocol Violation | 1
Not completed — Missing discontinuation information | 15

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1069
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was missing for 1 participant; therefore, the population for age included 1068 participants.
  years | 52.21 (10.70)
Sex/Gender, Customized [Number; unit: participants]
  Female | 472
  Male | 589
  Missing | 8
Region of Enrollment [Number; unit: participants]
  India | 1069

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between HbA1c Values at Week 12 and Hypoglycemia Scores
Description: Coefficient of correlation was measured using a linear regression analysis for the association between two variables, HbA1c values at Week 12 and hypoglycemia scores. A negative correlation coefficient indicates that as one value increases the other value decreases, and vice versa.
Time Frame: Week 12
Population: Evaluable population defined as all enrolled participants who completed the study and had the values for HbA1c at Week 12 and Stanford Hypoglycemia Score without any major protocol deviation.
Measure: Number (95% Confidence Interval); unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 950
Correlation coefficient | -0.1215 (1.90) [-0.1836 to -0.0583]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority or Other; p = 0.0002, Regression, Linear; Pearson correlation coefficient

2. Secondary Outcome: Hypoglycemia Symptom Score by Sub-group (Demographic/Disease Parameters)
Description: Sub-group analyses of mean hypoglycemia symptom score. Participants were grouped based on gender, age, hypoglycemia severity, body mass index, duration of diabetes, and number of oral hypoglycemic agents. Hypoglycemia symptom score (measured by Stanford Hypoglycemia Questionnaire) is a score on a scale with a possible range of 0 (best) to 7 (worst). The questionnaire was administered by the physician at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 950
Score on a scale
  Male, n=526 | 0.87 (1.37)
  Female, n=417 | 1.12 (1.46)
  Age 18-34 years, n=45 | 0.91 (1.62)
  Age 35-44 years, n=171 | 0.87 (1.36)
  Age 45-64 years, n=595 | 0.96 (1.39)
  Age 65 years and older, n=138 | 1.18 (1.49)
  Mild hypoglycemia, n=286 | 1.59 (1.38)
  Moderate hypoglycemia, n=168 | 2.36 (1.49)
  Severe hypoglycemia, n=15 | 2.53 (1.68)
  Body mass index <25 kg/m^2, n=370 | 1.01 (1.44)
  Body mass index 25-30 kg/m^2, n=394 | 0.95 (1.42)
  Body mass index >30 kg/m^2, n=183 | 0.96 (1.37)
  Duration of T2DM <5 years, n=640 | 0.88 (1.36)
  Duration of T2DM 5-10 years, n=239 | 1.15 (1.52)
  Duration of T2DM >10 years, n=49 | 1.29 (1.46)
  No background oral hypoglycemic agents, n=20 | 0.60 (0.99)
  1 background oral hypoglycemic agent, n=854 | 0.97 (1.41)
  2 background oral hypoglycemic agents, n=69 | 1.30 (1.61)
  3 background oral hypoglycemic agents, n=7 | 0.00 (0.00)

3. Secondary Outcome: Correlation Between HbA1c Values at Week 12 and Hypoglycemia Scores by Sub-group (Demographic/Disease Parameters)
Description: Sub-group analyses based on Karl pearson coefficient of correlation for HbA1c values at Week 12 and hypoglycemia score. Participants were grouped based on gender, age, body mass index, and duration of diabetes. A negative correlation coefficient indicates that as one value increases the other value decreases, and vice versa.
Time Frame: Week 12
Measure: Number; unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 950
Correlation coefficient
  Male, n=526 | -0.1654
  Female, n=417 | -0.0756
  Age 18-34 years, n=45 | -0.1636
  Age 35-44 years, n=171 | -0.1034
  Age 45-64 years, n=595 | -0.1222
  Age 65 years and older, n=138 | -0.0984
  Body mass index <25 kg/m^2, n=370 | -0.0100
  Body mass index 25-30 kg/m^2, n=394 | -0.2188
  Body mass index >30 kg/m^2, n=183 | -0.1688
  Duration of diabetes <5 years, n=640 | -0.1201
  Duration of diabetes 5-10 years, n=239 | -0.1503
  Duration of diabetes >10 years, n=49 | -0.1316

4. Secondary Outcome: Correlation Between HbA1c Values at Baseline and Hypoglycemia Scores at Week 12
Description: Coefficient of correlation as measured using linear regression analysis for association between two variables, HbA1c values at baseline and hypoglycemia scores. A positive correlation coefficient indicates that as one value increases the other value increases, or as as one value decreases the other value decreases.
Time Frame: Baseline and Week 12
Population: All enrolled participants with available data at both Baseline and Week 12.
Measure: Number; unit: Correlation coefficient
Arm/Group | All Participants
Number analyzed (Participants) | 899
Correlation coefficient | 0.0026

ADVERSE EVENTS:
Description: No adverse events were recorded separately other than hypoglycemia.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/1069
Other Adverse Events (participants affected / at risk) | 492/1069
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1069)
Hypoglycemia (Metabolism and nutrition disorders) | 492 (2968)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the study sponsor as confidential must be deleted prior to submission.